CLINICAL TRIAL: NCT03795974
Title: Evaluation of the Efficacy of Allogeneic Umbilical Cord Derived Hematopoietic Stem Cells and Mesenchymal Stromal Cells in Patients With Spastic Cerebral Palsy on Developmental Function , A Clinical Trial phase2
Brief Title: Efficacy of Allogeneic Umbilical Cord Derived Hematopoietic and Mesenchymal Stem Cells in Cerebral Palsy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Hormozgan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Mahmoud Reza Ashrafi, Professor of Pediatric Neurology, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRCT201706176907N13
Record Dates: First submitted 2018-12-03; First posted 2019-01-08 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2019-01

CONDITIONS: Cerebral Palsy, Spastic
Keywords: Quadriparetic CP, Diparetic CP, Spastic
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Intervention Model Description: HLA typing were done for 150 cases of spastic CP with our inclusion criteria and 36 cases of class 6 matching of HLA selected for hematopoietic stem cells derived from allogenic umbilical cord and 72 cases were randomly divided to Mesenchymal cells derived from allogenic umbilical cord and control group .
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: only one of the investigators knows the type of cell therapy for intervention group and simulation of intrathecal injection for control group .
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MNC & MSC with Control (Active Comparator): One intrathecal injection of Hematopoietic stem cells and Mesenchymal stem cells derived from allogenic umbilical cord for each group of 36 cases of spastic CP and neurorehabilitation during the 12 months of follow up of clinical evaluation of developmental functions and spasticity
  Interventions: Biological: MNC; Biological: MSC; Procedure: Control
- MNC & MSC (Experimental): Comparison of effects of intrathecal injection of MNC and MSC on improvement of developmental functions and spasticity of CP patients
  Interventions: Biological: MNC; Biological: MSC

INTERVENTIONS:
Biological: MNC — Hematopoietic stem cells derived from allogenic umbilical cord
  Other Names: Hematopoietic stem cells
Biological: MSC — Mesenchymal cells derived from allogenic umbilical cord
  Other Names: Mesenchymal stem cells
Procedure: Control — control group without injection and appearance simulating lumbar puncture without awareness of the patients and evaluators , but rehabilitation continued .
  Arms: MNC & MSC with Control

SUMMARY:
Cerebral palsy(CP) consisted of a group of developmental disability in the field of motor function and is one of the major problems of pediatric neurology and at the present time there is no standard curative medical or surgical treatment for it .Stem cell therapy is one of a new and hopeful therapeutic methods of therapy for CP .This double blind study designed for the evaluation of safety and therapeutic effects of intrathecal hematopoietic and mesenchymal stem cells derived from allogenic umbilical cord in change and probable improvement of developmental functions of spastic CP participants between 4-14 years old and comparing with control group of CP participants without cell therapy . 108 cases recruited and randomly divided to 3 groups of 36 cases : hematopoietic stem cells derived from allogenic umbilical cord , Mesenchymal cells derived from allogenic umbilical cord and control group without injection and appearance simulating lumbar puncture without awareness of the patients and evaluators . Developmental functions and spasticity evaluated before intervention and will be done 1 , 3 , 6 and 12 months after injection . During this period neuro rehabilitation will be continued . Brain neuroimaging were done at the recruitment time and will be repeated after 12 months .

DETAILED DESCRIPTION:
CP is characterized by aberrant control of movement or posture of a patient , appearing early in life , and not the result of a recognized progressive or degenerative brain disease . CP is an umbrella term and represents a group of conditions (not a single disorder) , has a broad range of expression with a static condition originally within the developing central nervous system . CP Is a disturbance of movement and or posture . At the present time there is no standard medical or surgical treatment for it .Stem cell therapy is a new and promising treatment .

150 cases of diparetic and quadiparetic spastic CP between 4-14 years old selected among the patients referred to the pediatric neurology outpatient department of Children's Medical Center Hospital (CMC) affiliated to Tehran University of Medical Sciences and had our inclusion criteria. HLA analysis were done for these patients and 36 cases of class 6 matched cases enrolled to the hematopoietic stem cells derived from allogenic umbilical cord (MNC) because of necessity of Human Leukocyte Antigen (HLA) matching in this type of cells and 72 cases among the remaining patients randomly divided to Mesenchymal stem cells derived from allogenic umbilical cord (MSC) and control group . Therefore 108 cases enrolled in 3 divided group of 36 patients .

Patients admitted to CMC hospital and intrathecal injection were done with sedation . Only one injection of stem cell was done for each patient . In the control group after insertion of the needle into the skin with an appearance of lumbar puncture simulation , no injection were done without the awareness of the patients or their parents. All of the patients admitted for one day and discharged the next day . As we wrote in the consent form for ethical consideration we are committed to perform stem cell injection for control participants free of charge after 12 months of the follow up . All of the participants will be referred for neurorehabilitation with a identical protocol .Both parents and clinical evaluators are not aware of the 3 divided groups and our study is double blind .Outcome measures will be evaluated 1, 3, 6. and 12 months after intervention .

Standard brain Magnetic Resonance Imaging (MRI) with Magnetic Resonance Spectroscopy (MRS) and Diffusion Tensor Imaging (DTI) were done before injection as baseline and will be repeated after 12 months of clinical follow up . This study designed for the evaluation of therapeutic effects of intrathecal MNC and MSC derived from allogenic umbilical cord in change and probable improvement of developmental functions of spastic CP patients between 4-14 years old in comparison with control group .Different scoring systems such as Gross Motor Functional Classification System (GMFCS) , Gross Motor Function Measure Score (GMFM66) , Manual Ability Classification System (MACS) , Pediatric Evaluation of Disability Inventory (PEDI) , CP QOL , Life Habits Questionnaire and Modified Ashworth scale for spasticity were done at baseline and then will be repeated in follow ups until 12 months of final evaluation .

Acute side effects and probable long term side effects will be reported and noted on our preformed questioners .

ELIGIBILITY:
Inclusion criteria :

* Spastic cerebral palsy (Diparetic , Quadriparetic)
* Ages between 4 - 14 years
* Gross motor function classification ( GMFC) between 2 -5
* No seizure disorder or with controlled seizures
* Evidence of definite acquired abnormal imaging findings compatible with CP
* Informed consent is taken from their parents

Exclusion criteria:

* Normal brain MRI
* Progressive neurologic disorders
* Congenital cortical malformations
* TORCH infections (Toxoplasmosis,Other,Rubella,Cytomegalovirus and Herpes infections)
* Other types of cerebral palsy including athetoid , atonic , ataxic , and mixed type
* Acute intercurrent infections such as Hepatitis C Virus (HCV), Hepatitis B Virus (HBV), Human Immunodeficiency Virus (HIV) Malignancies
* Hemorrhagic diathesis
* Severe anemia ( Hemoglobin less than 8 g/dl )
* Ventilator dependent pulmonary diseases
* Renal insufficiency
* Severe liver dysfunction

Ages: 4 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2017-07-23 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline Gross Motor Function Classification System (GMFCS) | Baseline
  The Gross Motor Function Classification System (GMFCS) for cerebral palsy is based on self-initiated movement, with emphasis on sitting, transfers, and mobility. When defining a five-level classification system, our primary criterion has been that the distinctions between levels must be meaningful in daily life. Distinctions are based on functional limitations, the need for hand-held mobility devices (such as walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement.
  LEVEL I - Walks without Limitations LEVEL II - Walks with Limitations LEVEL III - Walks Using a Hand-Held Mobility Device LEVEL IV - Self-Mobility with Limitations; May Use Powered Mobility LEVEL V - Transported in a Manual Wheelchair We enrolled the patients with GMFCS more than class II and evaluate for change of this scale during the follow up period . Lower scores demonstrate better gross motor function of children .
Change from baseline Gross Motor Function Classification System (GMFCS) | "month" 3
  The Gross Motor Function Classification System (GMFCS) for cerebral palsy is based on self-initiated movement, with emphasis on sitting, transfers, and mobility. When defining a five-level classification system, our primary criterion has been that the distinctions between levels must be meaningful in daily life. Distinctions are based on functional limitations, the need for hand-held mobility devices (such as walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement.
  LEVEL I - Walks without Limitations LEVEL II - Walks with Limitations LEVEL III - Walks Using a Hand-Held Mobility Device LEVEL IV - Self-Mobility with Limitations; May Use Powered Mobility LEVEL V - Transported in a Manual Wheelchair We enrolled the patients with GMFCS more than class II and evaluate for change of this scale during the follow up period . Lower scores demonstrate better gross motor function of children .
Change from baseline Gross Motor Function Classification System (GMFCS) | "month" 6
  The Gross Motor Function Classification System (GMFCS) for cerebral palsy is based on self-initiated movement, with emphasis on sitting, transfers, and mobility. When defining a five-level classification system, our primary criterion has been that the distinctions between levels must be meaningful in daily life. Distinctions are based on functional limitations, the need for hand-held mobility devices (such as walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement.
  LEVEL I - Walks without Limitations LEVEL II - Walks with Limitations LEVEL III - Walks Using a Hand-Held Mobility Device LEVEL IV - Self-Mobility with Limitations; May Use Powered Mobility LEVEL V - Transported in a Manual Wheelchair We enrolled the patients with GMFCS more than class II and evaluate for change of this scale during the follow up period . Lower scores demonstrate better gross motor function of children .
Change from baseline Gross Motor Function Classification System (GMFCS) | "month" 12
  The Gross Motor Function Classification System (GMFCS) for cerebral palsy is based on self-initiated movement, with emphasis on sitting, transfers, and mobility. When defining a five-level classification system, our primary criterion has been that the distinctions between levels must be meaningful in daily life. Distinctions are based on functional limitations, the need for hand-held mobility devices (such as walkers, crutches, or canes) or wheeled mobility, and to a much lesser extent, quality of movement.
  LEVEL I - Walks without Limitations LEVEL II - Walks with Limitations LEVEL III - Walks Using a Hand-Held Mobility Device LEVEL IV - Self-Mobility with Limitations; May Use Powered Mobility LEVEL V - Transported in a Manual Wheelchair We enrolled the patients with GMFCS more than class II and evaluate for change of this scale during the follow up period . Lower scores demonstrate better gross motor function of children .
Change from baseline GROSS MOTOR FUNCTION MEASURE (GMFM66) | Baseline
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy.
  GMFM 66 contained 66 item and each item include 4 score (0-3) SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes We are using validated Persian version of GMFM 66 in this research. Higher scores demonstrate better gross motor function of children.
Change from baseline GROSS MOTOR FUNCTION MEASURE (GMFM66) | "month" 1
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy.
  GMFM 66 contained 66 item and each item include 4 score (0-3) SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes We are using validated Persian version of GMFM 66 in this research. Higher scores demonstrate better gross motor function of children.
Change from baseline GROSS MOTOR FUNCTION MEASURE (GMFM66) | "month" 3
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy.
  GMFM 66 contained 66 item and each item include 4 score (0-3) SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes We are using validated Persian version of GMFM 66 in this research. Higher scores demonstrate better gross motor function of children.
Change from baseline GROSS MOTOR FUNCTION MEASURE (GMFM66) | "month" 6
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy.
  GMFM 66 contained 66 item and each item include 4 score (0-3) SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes We are using validated Persian version of GMFM 66 in this research. Higher scores demonstrate better gross motor function of children.
Change from baseline GROSS MOTOR FUNCTION MEASURE (GMFM66) | "month" 12
  The GMFM is a standardized observational instrument designed and validated to measure change in gross motor function over time in children with cerebral palsy.
  GMFM 66 contained 66 item and each item include 4 score (0-3) SCORING KEY 0 = does not initiate 1 = initiates 2 = partially completes 3 = completes We are using validated Persian version of GMFM 66 in this research. Higher scores demonstrate better gross motor function of children.
Change from baseline Manual Ability Classification System for Children with Cerebral Palsy (MACS) | Baseline
  The Manual Ability Classification System (MACS)describes how children with cerebral palsy (CP)use their hands to handle objects in daily activities.
  MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.
  1. Handle objects easily and successfully
  2. Handles most objects but with somewhat reduced quality and/or speed of achievement
  3. Handle objects with difficulty; needs help to prepare and/or modify activities
  4. Handles a limited selection of easily managed objects in adapted situations
  5. Does not handle objects and has severely limited ability to perform even simple actions Level I include children with minor limitations, while children with severe functional limitations will usually be found at levels IV and V.
  We are using validated Persian classification system.
Change from baseline Manual Ability Classification System for Children with Cerebral Palsy (MACS) | "month" 3
  The Manual Ability Classification System (MACS)describes how children with cerebral palsy (CP)use their hands to handle objects in daily activities.
  MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.
  1. Handle objects easily and successfully
  2. Handles most objects but with somewhat reduced quality and/or speed of achievement
  3. Handle objects with difficulty; needs help to prepare and/or modify activities
  4. Handles a limited selection of easily managed objects in adapted situations
  5. Does not handle objects and has severely limited ability to perform even simple actions Level I include children with minor limitations, while children with severe functional limitations will usually be found at levels IV and V.
  We are using validated Persian classification system.
Change from baseline Manual Ability Classification System for Children with Cerebral Palsy (MACS) | "month" 6
  The Manual Ability Classification System (MACS)describes how children with cerebral palsy (CP)use their hands to handle objects in daily activities.
  MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.
  1. Handle objects easily and successfully
  2. Handles most objects but with somewhat reduced quality and/or speed of achievement
  3. Handle objects with difficulty; needs help to prepare and/or modify activities
  4. Handles a limited selection of easily managed objects in adapted situations
  5. Does not handle objects and has severely limited ability to perform even simple actions Level I include children with minor limitations, while children with severe functional limitations will usually be found at levels IV and V.
  We are using validated Persian classification system.
Change from baseline Manual Ability Classification System for Children with Cerebral Palsy (MACS) | "month" 12
  The Manual Ability Classification System (MACS)describes how children with cerebral palsy (CP)use their hands to handle objects in daily activities.
  MACS describes five levels. The levels are based on the children's self-initiated ability to handle objects and their need for assistance or adaptation to perform manual activities in everyday life.
  1. Handle objects easily and successfully
  2. Handles most objects but with somewhat reduced quality and/or speed of achievement
  3. Handle objects with difficulty; needs help to prepare and/or modify activities
  4. Handles a limited selection of easily managed objects in adapted situations
  5. Does not handle objects and has severely limited ability to perform even simple actions Level I include children with minor limitations, while children with severe functional limitations will usually be found at levels IV and V.
  We are using validated Persian classification system.
Change from baseline Pediatric Evaluation of Disability Inventory (PEDI) | Baseline
  The PEDI contains items to measure functional capability, and also items to measure the performance in three content domains: Self Care (SC), Mobility (M) and Social Function (SF), Capability is measured by the assessment of the functional skills of which the child has shown mastery.
  The items in the FSS are discrete and are accompanied by scoring criteria and sometimes examples of behavior to help clarify scoring decisions. The items can be scored 0 or 1. 0 = unable or limited in capability to perform item in most situations 1 = capable of performing item in most situations, or item has been previously mastered and functional skills have progressed beyond this level.
  We are using validated Persian version of this Questionnaire. Higher scores demonstrate better functional capability.
Change from baseline Pediatric Evaluation of Disability Inventory (PEDI) | "month" 6
  The PEDI contains items to measure functional capability, and also items to measure the performance in three content domains: Self Care (SC), Mobility (M) and Social Function (SF), Capability is measured by the assessment of the functional skills of which the child has shown mastery.
  The items in the FSS are discrete and are accompanied by scoring criteria and sometimes examples of behavior to help clarify scoring decisions. The items can be scored 0 or 1. 0 = unable or limited in capability to perform item in most situations 1 = capable of performing item in most situations, or item has been previously mastered and functional skills have progressed beyond this level.
  We are using validated Persian version of this Questionnaire. Higher scores demonstrate better functional capability.
Change from baseline Pediatric Evaluation of Disability Inventory (PEDI) | "month" 12
  The PEDI contains items to measure functional capability, and also items to measure the performance in three content domains: Self Care (SC), Mobility (M) and Social Function (SF), Capability is measured by the assessment of the functional skills of which the child has shown mastery.
  The items in the FSS are discrete and are accompanied by scoring criteria and sometimes examples of behavior to help clarify scoring decisions. The items can be scored 0 or 1. 0 = unable or limited in capability to perform item in most situations 1 = capable of performing item in most situations, or item has been previously mastered and functional skills have progressed beyond this level.
  We are using validated Persian version of this Questionnaire. Higher scores demonstrate better functional capability.
Change from baseline Modified Ashworth scale | Baseline
  Scoring (taken from Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension ankle plantar flexion ,knee flexion ,hip flexion , wrist flexion , elbow flexion will be exam-ed by Modified Ashwotth scale and change in severity of spasticity
  ankle plantar flexion,knee flexion,hip flexion,wrist flexion,elbow flexion,Spasticity improvement of patients according to Modified Ashworth scale
Change from baseline Modified Ashworth scale | "month" 1
  Scoring (taken from Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension ankle plantar flexion ,knee flexion ,hip flexion , wrist flexion , elbow flexion will be exam-ed by Modified Ashwotth scale and change in severity of spasticity
  ankle plantar flexion,knee flexion,hip flexion,wrist flexion,elbow flexion,Spasticity improvement of patients according to Modified Ashworth scale
Change from baseline Modified Ashworth scale | "month" 3
  Scoring (taken from Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension ankle plantar flexion ,knee flexion ,hip flexion , wrist flexion , elbow flexion will be exam-ed by Modified Ashwotth scale and change in severity of spasticity
  ankle plantar flexion,knee flexion,hip flexion,wrist flexion,elbow flexion,Spasticity improvement of patients according to Modified Ashworth scale
Change from baseline Modified Ashworth scale | "month" 6
  Scoring (taken from Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension ankle plantar flexion ,knee flexion ,hip flexion , wrist flexion , elbow flexion will be exam-ed by Modified Ashwotth scale and change in severity of spasticity
  ankle plantar flexion,knee flexion,hip flexion,wrist flexion,elbow flexion,Spasticity improvement of patients according to Modified Ashworth scale
Change from baseline Modified Ashworth scale | "month" 12
  Scoring (taken from Bohannon and Smith, 1987):
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension ankle plantar flexion ,knee flexion ,hip flexion , wrist flexion , elbow flexion will be exam-ed by Modified Ashwotth scale and change in severity of spasticity
  ankle plantar flexion,knee flexion,hip flexion,wrist flexion,elbow flexion,Spasticity improvement of patients according to Modified Ashworth scale

SECONDARY OUTCOMES:
Change from baseline acquired Brain Magnetic Resonance Imaging (MRI) findings | Baseline
  One of our inclusion criteria for enrollment of the cases was evidence of definite acquired abnormal imaging findings compatible with CP such as periventricular leukomalacia (PVL) , cystic encephalomalacia ,periventricular gliosis , porencephalic cyst , basal ganglia involvement and brain atrophy . Decrements in size or improvement of Brain imaging findings would be expected due to Stem Cell therapy and will be followed 12 months after injection .
Change from baseline acquired Brain Magnetic Resonance Imaging (MRI) findings | "month" 12
  One of our inclusion criteria for enrollment of the cases was evidence of definite acquired abnormal imaging findings compatible with CP such as periventricular leukomalacia (PVL) , cystic encephalomalacia ,periventricular gliosis , porencephalic cyst , basal ganglia involvement and brain atrophy . Decrements in size or improvement of Brain imaging findings would be expected due to Stem Cell therapy and will be followed 12 months after injection .
Change from baseline Brain Magnetic Resonance Spectroscopy (MRS) | Baseline
  MRS allows noninvasive detection and measurement of normal and abnormal metabolites and biochemical changes in the brain . The frequency of different metabolites is measured in units called parts per million (PPM) and plotted on a graph as peaks of varying height . The metabolites normally detected in the brain, regardless of the adopted echo time, include Nacetyl aspartate (NAA),a neuronal marker, choline (Cho), a membrane marker, and creatine (Cr), an energy metabolism marker. Increase in NAA /Cr and NAA/Cho ratios expected as baseline and would be expected to have a change after Stem Cell therapy in favor of neuroglia cells load or number increase at the site of previous brain damage.
Change from baseline Brain Magnetic Resonance Spectroscopy (MRS) | "month" 12
  MRS allows noninvasive detection and measurement of normal and abnormal metabolites and biochemical changes in the brain . The frequency of different metabolites is measured in units called parts per million (PPM) and plotted on a graph as peaks of varying height . The metabolites normally detected in the brain, regardless of the adopted echo time, include Nacetyl aspartate (NAA),a neuronal marker, choline (Cho), a membrane marker, and creatine (Cr), an energy metabolism marker. Increase in NAA /Cr and NAA/Cho ratios expected as baseline and would be expected to have a change after Stem Cell therapy in favor of neuroglia cells load or number increase at the site of previous brain damage.
Change from baseline Diffuse Tensor Imaging (DTI) fiber count of periventricular white matter | Baseline
  DTI is a modiﬁcation of the MRI technique that is sensitive to the Brownian motion of water molecules in biological tissues and is a new clinical method that can demonstrate the orientation and integrity of white matter ﬁbers . Periventricular white matter injury is a major form of brain injury observed in CP . Signiﬁcant reduction in DTI ﬁber count on the periventricular or other regions of cerebral white matter injury involving corticospinal tract , corticobulbar tract and superior thalamic radiation expected as baseline . Increase in DTI ﬁber count would be expected due to Stem Cell therapy and will be followed 12 months after injection .
Change from baseline Diffuse Tensor Imaging (DTI) fiber count of periventricular white matter | "month" 12
  DTI is a modiﬁcation of the MRI technique that is sensitive to the Brownian motion of water molecules in biological tissues and is a new clinical method that can demonstrate the orientation and integrity of white matter ﬁbers . Periventricular white matter injury is a major form of brain injury observed in CP . Signiﬁcant reduction in DTI ﬁber count on the periventricular or other regions of cerebral white matter injury involving corticospinal tract , corticobulbar tract and superior thalamic radiation expected as baseline . Increase in DTI ﬁber count would be expected due to Stem Cell therapy and will be followed 12 months after injection .

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoudreza Ashrafi, MD, Principal Investigator — Tehran University of Medical Sciences, Children's Medical Center; Amirali Hamidieh, MD, Study Director — Tehran University of Medical Sciences , Children's Medical Center; Hadi Montazerlotfelahi, MD, Study Director — Alborz University of Medical Sciences; Anahita Majma, MD, Study Director — Tehran University of Medical Sciences Children's Medical Center; Masood Ghahvechi akbari, MD, Study Director — Tehran University of Medical Sciences ,Children's Medical Center; Ali Reza Moaeidi, MD, Study Director — Hormozgan University of Medical Sciences
Locations (4):
- Iran (4):
  - Tehran University of Medical Sciences , Growth and Development Research Center- Children's Medical Center, Tehran
  - Tehran University of Medical Sciences Chidren's Medical Center Radiology Department, Tehran
  - Tehran University of Medical Sciences, Department of Pediatric Neurology , Children's Medical Center, Tehran
  - ROYAN Stem Cell Technology Co, Tehran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Papadopoulos KI, Low SS, Aw TC, Chantarojanasiri T. Safety and feasibility of autologous umbilical cord blood transfusion in 2 toddlers with cerebral palsy and the role of low dose granulocyte-colony stimulating factor injections. Restor Neurol Neurosci. 2011;29(1):17-22. doi: 10.3233/RNN-2011-0572. PMID 21335665
- [Background] Feng M, Lu A, Gao H, Qian C, Zhang J, Lin T, Zhao Y. Safety of Allogeneic Umbilical Cord Blood Stem Cells Therapy in Patients with Severe Cerebral Palsy: A Retrospective Study. Stem Cells Int. 2015;2015:325652. doi: 10.1155/2015/325652. Epub 2015 Jul 8. PMID 26236347
- [Background] Thomas B, Eyssen M, Peeters R, Molenaers G, Van Hecke P, De Cock P, Sunaert S. Quantitative diffusion tensor imaging in cerebral palsy due to periventricular white matter injury. Brain. 2005 Nov;128(Pt 11):2562-77. doi: 10.1093/brain/awh600. Epub 2005 Jul 27. PMID 16049045
- [Result] Zali A, Arab L, Ashrafi F, Mardpour S, Niknejhadi M, Hedayati-Asl AA, Halimi-Asl A, Ommi D, Hosseini SE, Baharvand H, Aghdami N. Intrathecal injection of CD133-positive enriched bone marrow progenitor cells in children with cerebral palsy: feasibility and safety. Cytotherapy. 2015 Feb;17(2):232-41. doi: 10.1016/j.jcyt.2014.10.011. Epub 2014 Nov 1. PMID 25593079
- [Result] Bax M, Goldstein M, Rosenbaum P, Leviton A, Paneth N, Dan B, Jacobsson B, Damiano D; Executive Committee for the Definition of Cerebral Palsy. Proposed definition and classification of cerebral palsy, April 2005. Dev Med Child Neurol. 2005 Aug;47(8):571-6. doi: 10.1017/s001216220500112x. PMID 16108461
- [Result] Shevell MI, Dagenais L, Hall N; REPACQ CONSORTIUM*. The relationship of cerebral palsy subtype and functional motor impairment: a population-based study. Dev Med Child Neurol. 2009 Nov;51(11):872-7. doi: 10.1111/j.1469-8749.2009.03269.x. Epub 2009 Mar 11. PMID 19416339
- [Result] Ashwal S, Russman BS, Blasco PA, Miller G, Sandler A, Shevell M, Stevenson R; Quality Standards Subcommittee of the American Academy of Neurology; Practice Committee of the Child Neurology Society. Practice parameter: diagnostic assessment of the child with cerebral palsy [RETIRED]: report of the Quality Standards Subcommittee of the American Academy of Neurology and the Practice Committee of the Child Neurology Society. Neurology. 2004 Mar 23;62(6):851-63. doi: 10.1212/01.wnl.0000117981.35364.1b. PMID 15037681
- [Result] Wang X, Cheng H, Hua R, Yang J, Dai G, Zhang Z, Wang R, Qin C, An Y. Effects of bone marrow mesenchymal stromal cells on gross motor function measure scores of children with cerebral palsy: a preliminary clinical study. Cytotherapy. 2013 Dec;15(12):1549-62. doi: 10.1016/j.jcyt.2013.06.001. Epub 2013 Oct 5. PMID 24100132
- [Result] Romanov YA, Svintsitskaya VA, Smirnov VN. Searching for alternative sources of postnatal human mesenchymal stem cells: candidate MSC-like cells from umbilical cord. Stem Cells. 2003;21(1):105-10. doi: 10.1634/stemcells.21-1-105. PMID 12529557
- [Result] Crompton KE, Elwood N, Kirkland M, Clark P, Novak I, Reddihough D. Feasibility of trialling cord blood stem cell treatments for cerebral palsy in Australia. J Paediatr Child Health. 2014 Jul;50(7):540-4. doi: 10.1111/jpc.12618. Epub 2014 Jun 9. PMID 24909743
- [Derived] Zarrabi M, Akbari MG, Amanat M, Majmaa A, Moaiedi AR, Montazerlotfelahi H, Nouri M, Hamidieh AA, Badv RS, Karimi H, Rabbani A, Mohebbi A, Rahimi-Dehgolan S, Rahimi R, Dehghan E, Vosough M, Abroun S, Shamsabadi FM, Tavasoli AR, Alizadeh H, Pak N, Zamani GR, Mohammadi M, Javadzadeh M, Ghofrani M, Hassanpour SH, Heidari M, Taghdiri MM, Mohseni MJ, Noparast Z, Masoomi S, Goudarzi M, Mohamadpour M, Shodjaee R, Samimi S, Mohammad M, Gholami M, Vafaei N, Koochakzadeh L, Valizadeh A, Malamiri RA, Ashrafi MR. The safety and efficacy of umbilical cord blood mononuclear cells in individuals with spastic cerebral palsy: a randomized double-blind sham-controlled clinical trial. BMC Neurol. 2022 Mar 29;22(1):123. doi: 10.1186/s12883-022-02636-y. PMID 35351020
- [Derived] Amanat M, Majmaa A, Zarrabi M, Nouri M, Akbari MG, Moaiedi AR, Ghaemi O, Zamani F, Najafi S, Badv RS, Vosough M, Hamidieh AA, Salehi M, Montazerlotfelahi H, Tavasoli AR, Heidari M, Mohebi H, Fatemi A, Garakani A, Ashrafi MR. Clinical and imaging outcomes after intrathecal injection of umbilical cord tissue mesenchymal stem cells in cerebral palsy: a randomized double-blind sham-controlled clinical trial. Stem Cell Res Ther. 2021 Aug 6;12(1):439. doi: 10.1186/s13287-021-02513-4. PMID 34362453

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-18): https://cdn.clinicaltrials.gov/large-docs/74/NCT03795974/Prot_SAP_000.pdf